CLINICAL TRIAL: NCT02138526
Title: Improving the Tolerability of the Oral Targeted Anticancer Drug Pazopanib by Food Intake (DIET)
Brief Title: Pazopanib Tolerability When Given With Food
Acronym: DIET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF-13.05
Record Dates: First submitted 2014-04-29; First posted 2014-05-14 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: cancer; pazopanib; food; pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fasted (Active Comparator): Intake of pazopanib in agreement with drug label - fasted state
  Interventions: Drug: pazopanib
- Continental breakfast (Experimental): Intake of a reduced equivalent pazopanib dose with a continental breakfast
  Interventions: Drug: pazopanib; Other: continental breakfast

INTERVENTIONS:
Drug: pazopanib — pazopanib 800mg OD without food
  Other Names: Votrient
Other: continental breakfast — pazopanib 600mg OD with food
  Arms: Continental breakfast

SUMMARY:
Pazopanib (Votrient) is registered for the treatment of patients with advanced renal cell carcinoma and patients with soft tissue sarcoma who have received prior chemotherapy. It is administered at a fixed oral dose of 800 mg once daily (OD) regardless of size, age and clinical condition. It is absorbed from the gastrointestinal tract with an oral bioavailability of ~21%. Pazopanib is practically insoluble and highly permeable. When ingested with high fat food the pazopanib exposure (area under the concentration time curve (AUC)) is doubled. Common adverse effects are diarrhea and nausea. This might be caused by the non-absorbed proportion of pazopanib. A reduced dose taken with food could be a possible approach to reduce these side effects. Therefore the investigators initially want to determine the equivalent reduced dose of pazopanib when taken with a continental breakfast. Thereafter the investigators want to investigate whether the intake with food reduces the frequently reported side effects nausea and diarrhea.

DETAILED DESCRIPTION:
Pazopanib (Votrient) is a multi targeted tyrosine kinase inhibitor of vascular endothelial growth factor receptor, (VEGFR-1, -2 en -3), platelet-derived growth factor receptor (PDGFR-α and -β), and stem cell factor receptor (c-KIT). Pazopanib is registered for the treatment of patients with advanced renal cell carcinoma and patients with soft tissue sarcoma who have received prior chemotherapy. It is administered at a fixed oral dose of 800 mg OD regardless of size, age and clinical condition. It is absorbed from the gastrointestinal tract with an oral bioavailability of ~21%. Pazopanib is practically insoluble and highly permeable. When ingested with high fat food the pazopanib exposure (area under the concentration time curve (AUC)) is doubled. Common adverse effects are diarrhea and nausea. This might be caused by the non-absorbed proportion of pazopanib. A dose reduction when ingested with food could be a logical approach to reduce these side effects; however this is not tested in patients yet. Therefore we want to perform a bioequivalent study to investigate what dose with a continental breakfast equals the dose of 800 mg in fasted conditions (study part A). In part B of the study we want to investigate whether the intake with food reduces the frequently reported side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.

   Note: informed consent may be obtained prior to start of the specified screening window.

   Note: procedures conducted as part of the subject's routine clinical management (e.g. blood count) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
2. ≥ 18 year old men and women who use pazopanib
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Adequate organ system function

Exclusion Criteria:

1. Poorly controlled hypertension; systolic blood pressure (SBP) ≥ 40 mm Hg or diastolic blood pressure (DBP) ≥ 90 mm Hg.

   Note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement. These three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure. The mean SBP / DBP ratio must be <140/90 mmHg (OR 150/90 mm Hg, if this criterion is approved by Safety Review Team) in order for a subject to be eligible for the study.
2. Corrected QT interval (QTc) > 480msecs.
3. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
4. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with risk of bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation.
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
5. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   * Malabsorption syndrome.
   * Major resection of the stomach or small bowel.
6. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

   Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
7. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
8. Evidence of active bleeding or bleeding diathesis.
9. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.

   Note: Lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessel is acceptable (CT with contrast is strongly recommended to evaluate such lesions).
10. Recent hemoptysis (½ teaspoon of red blood within 8 weeks before first dose of study drug).
11. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
12. Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of day 1 and for the duration of the study.
13. Concurrent use of other substances known or likely to interfere with the pharmacokinetics of pazopanib.

    Patients, who are adjusted to proton pump inhibitors and had no dose modifications for over two weeks, are allowed to participate
14. Women of childbearing potential without adequate contraception, pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of pazopanib | 4 weeks
  Determination of AUC of pazopanib when taken with a continental breakfast compared to 800 mg in fasted state (geometric mean ratio will be determined)

SECONDARY OUTCOMES:
number of side effects | 2 months
  Number of side effects will be compared for the two treatments (with and food.
questionnaire | 2 months
  Preference of patients (by questionnaire): intake of pazopanib with or without

CONTACTS AND LOCATIONS:
Overall Officials: Nielka P. van Erp, PharmD, PhD, Principal Investigator — Department of Pharmacy, Radboudumc; Carla M.L. van Herpen, MD, PhD, Principal Investigator — Department of Medical Oncology, Radboudumc
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Lubberman FJE, Gelderblom H, Hamberg P, Vervenne WL, Mulder SF, Jansman FGA, Colbers A, van der Graaf WTA, Burger DM, Luelmo S, Moes DJAR, van Herpen CML, van Erp NP. The Effect of Using Pazopanib With Food vs. Fasted on Pharmacokinetics, Patient Safety, and Preference (DIET Study). Clin Pharmacol Ther. 2019 Nov;106(5):1076-1082. doi: 10.1002/cpt.1515. Epub 2019 Jul 9. PMID 31125423
- [Derived] Krens SD, Lubberman FJE, van Egmond M, Jansman FGA, Burger DM, Hamberg P, Vervenne WL, Gelderblom H, van der Graaf WTA, Desar IME, van Herpen CML, van Erp NP. The impact of a 1-hour time interval between pazopanib and subsequent intake of gastric acid suppressants on pazopanib exposure. Int J Cancer. 2021 Jun 1;148(11):2799-2806. doi: 10.1002/ijc.33469. Epub 2021 Jan 19. PMID 33428771
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/31125423/